CLINICAL TRIAL: NCT04898413
Title: Group-based Acceptance and Commitment Therapy and Group-based Cognitive Behavior Therapy for Family Caregivers of People With Dementia in Japan
Brief Title: Group-based Acceptance and Commitment Therapy for Family Caregivers of People With Dementia in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meiji Gakuin University (Other)
Responsible Party: Principal Investigator, Hiroshi Morimoto, Associate professor, Meiji Gakuin University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MG21PS0401; 21K03094 (Other Grant/Funding Number: Japan Society for the Promotion of Science)
Record Dates: First submitted 2021-05-13; First posted 2021-05-24 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Family Caregivers
Keywords: Dementia; Family caregivers; Acceptance and commitment therapy; Cognitive behavior therapy; Reminiscence therapy
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-based acceptance and commitment therapy (ACT) (Experimental): Participants assigned to the group-based ACT intervention will receive eight sessions through face-to-face or Zoom video conferencing over the course of four months. Participants will also receive individualized support between sessions to help them better understand the program using phone or Zoom video conferencing. If participants' care recipient hopes to receive psychological treatment, they will be invited to participate in a group-based reminiscence therapy held once or twice a month, each lasting about 60-90 minutes, over the course of about three months.
  Interventions: Behavioral: Group-based acceptance and commitment therapy (ACT)
- Group-based cognitive behavior therapy (CBT) (Active Comparator): Participants assigned to the group-based CBT intervention will receive eight sessions through face-to-face or Zoom video conferencing over the course of four months. Participants will also receive individualized support between sessions to help them better understand the program using phone or Zoom video conferencing. If participants' care recipient hopes to receive psychological treatment, they will be invited to participate in a group-based reminiscence therapy held once or twice a month, each lasting about 60-90 minutes, over the course of about three months.
  Interventions: Behavioral: Group-based cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Group-based acceptance and commitment therapy (ACT) — Group-based ACT intervention by professional psychotherapist consists of four modules: (a) psychoeducation about dementia and experiential avoidance in caregiving, (b)mindfulness and acceptance of aversive emotions, sensations, and thoughts, (c) behavior management for care recipients' BPSD, and (d) clarifying and choosing one's value, and taking actions toward the chosen values. Each session lasts about 90 minutes and will be held every two weeks. Group-based reminiscence therapy for care recipients will be conducted by a professional psychotherapist other than the one conducting group-based ACT intervention.
  Arms: Group-based acceptance and commitment therapy (ACT)
Behavioral: Group-based cognitive behavioral therapy (CBT) — Group-based CBT intervention by professional psychotherapist consists of four modules: (a) psychoeducation about dementia and distress in caregiving, (b) cognitive restructuring and relaxation, (c) behavior management for care recipients' BPSD, and (d) increasing pleasant activities. Each session lasts about 90 minutes and will be held every two weeks. Group-based reminiscence therapy for care recipients will be conducted by a professional psychotherapist other than the one conducting group-based CBT intervention.
  Arms: Group-based cognitive behavior therapy (CBT)

SUMMARY:
Along with more people worldwide having dementia, the number of people with dementia and their family caregivers have increased in Japan. However, psychological support for family caregivers of people with dementia is still limited in Japan. The purpose of this pilot study is to examine feasibility and preliminary efficacy of a group-based acceptance and commitment therapy (ACT) for family caregivers of people with dementia in Japan compared to a group-based cognitive behavior therapy (CBT). This study also preliminarily examines the efficacy of combining psychological intervention for family caregivers (group-based ACT/CBT) with psychological intervention for their care recipients (group-based reminiscence therapy).

DETAILED DESCRIPTION:
This study employs quasi-experimental design to investigate the feasibility and preliminary efficacy of the group-based ACT for family caregivers of people with dementia compared to the group-based CBT. Both interventions consist of eight sessions, each lasting about 90 minutes, through face-to-face or Zoom video conferencing over the course of four months. Family caregivers will be assigned to either the ACT or CBT interventions. Pre-, post-intervention, and 6 month follow-up measurements assess depression, anxiety, quality of life, cognitive appraisal of caregiving (i.e., subjective burden and positive aspect of caregiving), possible process factors (i.e., caregiving self-efficacy, experiential avoidance, and commitment), care recipients' behavioral and psychological symptoms of dementia (BPSD), and so on. This study also preliminarily examines the efficacy of combining psychological intervention for family caregivers (i.e., the group-based ACT/CBT) with those for their care recipients (i.e., group-based reminiscence therapy). The group-based reminiscence therapy will be held once or twice a month, each lasting about 60-90 minutes, over the course of about three months.

ELIGIBILITY:
Inclusion Criteria:

Family caregivers:

* providing care for a family member with dementia or mild cognitive impairment
* being able to speak and read Japanese
* being 20 years of age or older.

Care recipients (group-based reminiscence therapy):

* having a clear intention to participate in the intervention
* being able to speak Japanese
* being diagnosed with mild cognitive impairment or mild stage of dementia and MoCA scores ≥ 11
* obtaining consent from their family caregiver and their doctor to participate in the intervention.

Exclusion Criteria:

Family caregivers:

* having psychiatric disorder at the time of participation in the intervention.

Care recipients (group-based reminiscence therapy):

* having insufficient capacity to give consent to participate in the intervention
* being diagnosed with moderate to severe stage of dementia or MoCA scores < 11.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline depression and anxiety at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the Hospital Anxiety and Depression Scale. This scale comprises two seven-item subscales: depression and anxiety. Scale scores range from 0 to 21 for each subscale, where higher scores indicate worse outcome.
Change from baseline quality of life (QOL) at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the WHOQOL26. This scale comprises 26 items on four subscales: physical domain, psychological domain, social relationships, environment, and general health/QOL. Scale scores range from 7 to 35 for physical domain, 6 to 30 for psychological domain, 3 to 15 for social relationships, 8 to 40 for environment, and 2 to 10 for general health/QOL. Higher scores indicate better outcome.

SECONDARY OUTCOMES:
Change from baseline subjective burden at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the Zarit Burden Interview. This scale comprises 22 items, ranging from 0 to 88. Higher scores indicate worse outcome.
Change from baseline positive aspects of caregiving at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the Cognitive Caregiving Appraisal Scale. This scale comprises 26 items on three negative appraisal subscales (feelings of restriction of social life, anxiety about continuing caregiving, and distress of the relationships with others) and three positive appraisal subscales (fulfillment of caregiving roles, affection toward the caretakers, and self-growth by caregiving). Positive appraisal subscales are used. Scale scores range from 6 to 24 for fulfillment of caregiving roles, 4 to 16 for affection toward the caretakers, and 3 to 12 for self-growth by caregiving. Higher scores indicate better outcome.
Change from baseline caregiving self-efficacy at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the Revised Scale for Caregiving Self-efficacy. This scale comprises 15 items on three subscales: obtaining respite, responding to disruptive behaviors, and controlling upsetting thoughts. Scale scores range from 0 to 100 for each subscale, where higher scores indicate better outcome.
Change from baseline experiential avoidance in caregiving at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the Experiential Avoidance in Caregiving Questionnaire. This scale comprises 15 items on three subscales: active avoidant behaviors, intolerance of negative thoughts and emotions, and apprehension concerning negative internal experiences related to caregiving. Scale scores range from 6 to 30 for active avoidant behaviors, 4 to 16 for intolerance of negative thoughts and emotions, and 5 to 25 for apprehension concerning negative internal experiences related to caregiving. Higher scores indicate worse outcome.
Change from baseline commitment to values at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the Values Questionnaire. This scale comprises 10 items on two subscales: obstruction and progress. Scale scores range from 0 to 30 for each subscale. Higher scores for the obstruction indicate lower commitment (i.e., worse outcome), and higher scores for the progress indicate higher commitment (i.e., better outcome).
Change from baseline care recipients' behavioral and psychological symptoms of dementia (BPSD) at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the Neuropsychiatric Inventory Questionnaire. This scale comprises 12 items measuring various BPSD. Participants (i.e., family caregivers) rated state of their care recipient. Scale scores range from 0 to 60, where higher scores indicate worse outcome.

OTHER OUTCOMES:
Change from baseline caregiving demands at 4 and 10 months | Baseline (pre-intervention), 4 months (immediately after the intervention), and 10 months (6 month follow-up)
  Measured by the Caregiver Burden Scale. This scale comprises 26 items on seven subscales measuring support for care recipient's activities of daily living, burden of behavioral and psychological symptoms, concern about future caregiving burden, lack of informal support, lack of formal support, caregiving interference with other roles, and financial burden of caregiving. Higher scores indicate worse outcome.
Usability of the intervention | Immediately after the intervention
  Measured by 10 items. Scale scores range from 10 to 50, where higher scores indicate higher levels of perceived usability of the intervention (i.e., better outcome).
Change from baseline care recipient's cognitive function at 3 and 6 months | Baseline, 3 months (immediately after the intervention), 6 months (3 month follow-up)
  Measured by the Montreal Cognitive Assessment. This instrument is a cognitive screening test for the detection of mild cognitive impairment and Alzheimer's disease. Scale scores range from 0 to 30, where higher scores indicate better outcome. This test will be used for participants in the care recipient's program (i.e., group-based reminiscence therapy) in both face-to-face and online settings.
Change from baseline care recipient's depression at 3 and 6 months | Baseline, 3 months (immediately after the intervention), 6 months (3 month follow-up)
  Measured by the Japanese version of the Geriatric Depression Scale Short Version. This scale comprises 15 items, ranging from 0 to 15. Higher scores indicate worse outcome. This scale will be used for participants in the care recipient's program (i.e., group-based reminiscence therapy) in both face-to-face and online settings.
Change from baseline care recipient's psychological distress at 3 and 6 months | Baseline, 3 months (immediately after the intervention), 6 months (3 month follow-up)
  Measured by the Stress Response Scale. This scale comprises 18 items on three subscales: depression/anxiety, irritability/anger, and helplessness. Scale scores range from 0 to 18 for each subscale. Higher scores indicate worse outcome. This scale will be used for participants in the care recipient's program (i.e., group-based reminiscence therapy) in both face-to-face and online settings.
Baseline care recipient's cognitive function | Baseline
  Measured by the Mini-Mental State Examination. This instrument is a cognitive screening test for the detection of dementia. Scale scores range from 0 to 30, where higher scores indicate better outcome. This test will be used for participants in the care recipient's program (i.e., group-based reminiscence therapy) in the case of a face-to-face setting.
Baseline care recipient's cognitive function | Baseline
  Measured by the Hasegawa Dementia Scale-Revised. This instrument is a cognitive screening test for the detection of dementia. Scale scores range from 0 to 30, where higher scores indicate better outcome. This test will be used for participants in the care recipient's program (i.e., group-based reminiscence therapy) in the case of an online setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Meiji Gakuin University, Minato-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No